CLINICAL TRIAL: NCT06063369
Title: Palmitoylethanolamide (PEA) vs Placebo for Major Depression: a Phase II Exploratory Study
Brief Title: PEA vs. Placebo for Major Depression
Acronym: PEA-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Israeli Medical Center for Alzheimer's (Other)
Responsible Party: Principal Investigator, Prof Mark Weiser, Head Psychiatrist, The Israeli Medical Center for Alzheimer's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PEA-01
Record Dates: First submitted 2023-03-23; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Bipolar Depression; Major Depressive Disorder
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major | interventions — palmidrol

STUDY DESIGN:
Intervention Model Description: Phase II - Randomized, double blind, placebo-controlled, parallel group clinical trial.
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Palmitoylethanolamide 1200 mg (Experimental): Dose: PEA 1200 mg given in 300 mg capsules (2 capsules twice daily) Route of administration: oral Duration and frequency: study medication will be provided to patients in bottles every two weeks for the duration of the study (three dispensations).
  Formulation: PEA Dosing scheme: Patients will be instructed to take two capsules twice daily for the 42 days of the study.
  Interventions: Drug: Palmitoylethanolamide
- Matching placebo (Placebo Comparator): 2 capsules twice daily identical to study arm. Route of administration: oral Duration and frequency: pills will be provided to patients in bottles every two weeks for the duration of the study (three dispensations).
  Formulation: placebo in identical capsules. Dosing scheme: Patients will be instructed to take two capsules twice daily for the 42 days of the study.
  Interventions: Drug: Palmitoylethanolamide

INTERVENTIONS:
Drug: Palmitoylethanolamide — Dose: PEA 1200 mg given in 400 mg capsules (3 capsules per day) or Placebo Route of administration: oral Duration and frequency: study medication will be provided to patients in bottles every two weeks for the duration of the study (three dispensations).
  Formulation: PEA and placebo in identical capsules. Dosing scheme: Patients will be instructed to take two capsules twice daily for the 42 days of the study.
  Other Names: PEA

SUMMARY:
Major Depression is often resistant to treatment, and all of the currently marketed anti-depressants can cause significant side effects and may precipitate mania. The aim of this proposal is to perform a proof-of-concept RCT testing Palmitoylethanolamide (PEA) as a treatment for unipolar or bipolar depression, randomizing 100 patients to 6-week treatment with PEA 1200 mg/d or matching placebo. There are several rationales for this study: (A) PEA acts at the peroxisome proliferator-activated receptor-alpha (PPAR-α), stimulating Allo biosynthesis. Allo is an endogenous, positive allosteric modulator of GABA-A receptors in glutamatergic neurons, including cortical and hippocampal pyramidal glutamatergic neurons and may be one of the endogenous regulators of depression and anxiety. (B) Sage Therapeutics has developed Allo which is FDA approved to treat post-partum depression, and is testing a molecular modification which can be administered orally for post-partum depression and unipolar depression, with mixed efficacy results. Pregnenolone, a precursor of neurosteroids, has also been reported to improve bipolar depression. Based on animal models, PEA increases Allo synthesis in areas of the brain thought to be involved in anxiety and depression. It may also favor the biosynthesis of sulfated forms of Allo and congeners that inhibit tonic rather than phasic NMDA-mediated excitatory neurotransmission. Showing that PEA-induced selective inhibition of tonic NMDA neurotransmission improves depression might enable development of steroid-based NMDA-inhibitor therapeutics. In addition, PEA-induced Allo upregulation potentiates GABA-A receptor-mediated inhibition. The NMDA and the GABAergic mechanisms may act in concert to improve behavioral outcomes. Since PEA increases Allo in the brain where it is endogenously formed, it might be more effective compared with exogenous administration, which is not site specific. There is evidence of a role of inflammation in depression; PEA has potent immunoregulatory and anti-inflammatory effects by directly activating PPAR-α, which has a protective role against neuroinflammation by inhibiting the signaling mediated by toll-like receptor 4.There is one published study which shows that PEA has an antidepressant effect in unipolar depression, 58 patients were randomized to receive 1200 mg/d of PEA or placebo added-on to citalopram, showing clinical improvements in patients receiving PEA.

DETAILED DESCRIPTION:
This is a multi-center, 6-week, randomized, double blind, placebo-controlled clinical trial of PEA vs. placebo in patients with unipolar or bipolar disorder who are currently in a Major Depressive Episode (MDE). PEA or placebo will be administered as monotherapy and any antidepressant, mood stabilizer or antipsychotic medication will be tapered down starting from the randomization day. The tapering process will be of one week, except for fluoxetine which will be tapered for a duration of two weeks.

At the screening visit, after signing the informed consent form, patients will be assessed using the MINI. MADRS and YMRS will be assessed for inclusion/exclusion criteria. Demographic information will be collected, psychiatric and medical history obtained, physical examination including height and weight, blood pressure and pulse rate will be performed. Blood samples for biochemistry analyses and CBC, and urine samples for urinalysis will be taken. Females of child-bearing potential will be tested for pregnancy. An ECG will be performed. Blood for neurosteroids and other biomarkers will be taken, processed to separate plasma from PBMC and stored, to be sent later to the laboratory of Dr. Pinna.

The baseline visit will be performed up to 7 days after screening. MADRS, CGI-BP/CGI-D, HAM-A and HAM-D will be collected. The use of concomitant medications as well as Adverse Events will be recorded throughout the study. Patients will be randomized to start study medication. The clinical questionnaires will be administered 2, 4 and 6 (End-of study, EOS) weeks after baseline. Biomarker analyses, including plasma neurosteroid and BDNF levels will be measured at baseline, and at the week 6 (EOS) visit. Concomitant medications and adverse events, as well as any other clinical change will be monitored through phone visits which will take place twice weekly on weeks 1, 3 and 5.

Study medication will be manufactured by Innexus Nutraceuticals in the Netherlands according to GMP, and will then be sent to Micronisierungs-Kontor Oberrot GmbH in Germany for micronization. The micronized compound will then be sent to PharmaMed Inc. in Pennsylvania, USA for packaging and labelling. Study medication will be randomized according to a computerized list supplied by the investigators to Innexus Nutraceuticals and PharmaMed Inc. Randomization of patients will be sequential. Kits will be kept in one central site, and after randomization patients from other site will be supplied with the kits.

Concomitant medication: After the screening visit, patients will start a tapering process for all antidepressant/antipsychotic/mood stabilizer. The tapering process will be of one week, except for fluoxetine which will be tapered for a duration of two weeks.

Rescue Medication: Up to 3 mg/day of lorazepam will be allowed as rescue medication in case of clinical deterioration, based on clinician's judgment.

Laboratory: Quantification of Allo and congeners, and PEA will performed by the state-of-the-art technology, GC-MS. The methodology to determine neurosteroid levels is a technique developed in Dr Pinna's lab (HPLC combined with GC-MS quantification), which allows the simultaneous determination of various neurosteroids from a single sample due to molar sensitivity and unsurpassed structural specificity.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM V criteria for a Major Depressive Episode, with or without a diagnosis of Bipolar I or Bipolar II disorder.
2. Between 18-65 years of age, male or female subjects of any race.
3. Able to provide informed consent. All participant patients must have signed an informed consent document indicating they understand the purpose of the study and are willing to complying with the study procedures and restrictions.
4. Have a MADRS above 20 and an YMRS < 12.
5. Inpatients or outpatients at the discretion of the investigator.
6. Live with a caregiver or have a relative/close friend who is in contact with them at least twice a week via phone.

Exclusion Criteria:

1. Diagnosis of schizophrenia or schizoaffective disorder
2. Women of child-bearing potential who do not practice contraception.
3. Women who are pregnant or breast-feeding.
4. Psychotic symptoms during the 2 weeks preceding the baseline day.
5. Failure of three or more antidepressant treatment trials.
6. Unstable medical disease (malignancy, poorly controlled diabetes, or cardiomyopathy, serious pulmonary disease, kidney disease, impaired liver functioning. Particular attention should be given to exclude patients with ischemic heart disease).
7. Has a clinically significant abnormal 12-lead electrocardiogram (ECG) at the Screening Visit, as determined by the Investigator.
8. At significant risk of committing suicide, or in the opinion of the Investigator, currently is at imminent risk of suicide or harming others.
9. Patients with a current DSM-V substance or alcohol dependence.
10. Concurrent delirium, mental retardation, drug-induced psychosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-12-21 (Estimated); Study Completion 2024-12-21 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D) | 6 weeks trial
  Depression Scale

SECONDARY OUTCOMES:
Clinical Global Impressions-Severity-Bipolar Scale or Clinical Global Impressions-Severity-Depression | 6 weeks trial
  Scale for Overall Bipolar Depression and Unipolar Depression severity
Hamilton Anxiety Rating Scale (HAM-A) | 6 weeks trial
  Anxiety Scake
Plasma measures including Allo and pregnanolone, their isomers, the sulfated congeners (pregnanolone sulphate and Allo sulphate) | 6 weeks trial
  neurosteroids
DHEA | 6 weeks trial
  measured with the state-of-the-art methodology gas chromatography mass spectrometry (GC-MS).
BDNF | 6 weeks trial
  Brain-derived neurotrophic factor
CRP | 6 weeks trial
  C-Reactive Protein
TLR-4 | 6 weeks trial
  Toll-like Receptor 4
Cytokines | 6 weeks trial
  Inflammatory markers

CONTACTS AND LOCATIONS:
Locations (1):
- State University of Medicine and Pharmacy " Nicolae Testemitsanu", Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No